CLINICAL TRIAL: NCT00003131
Title: A Study of the Efficacy and Safety of CMA-676 as Single Agent Treatment of Patients With Acute Myeloid Leukemia (AML) in First Relapse
Brief Title: CMA-676 in Treating Patients With Acute Myeloid Leukemia in First Relapse
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: W-AR-0903B1-201-US; CDR0000065896; UCCRC-8600; NCI-V97-1355
Record Dates: First submitted 1999-11-01; First posted 2004-08-24 (Estimated); Last update posted 2012-08-22 (Estimated); Status verified 2012-08

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — Drug Therapy; Gemtuzumab

INTERVENTIONS:
Drug: chemotherapy
Drug: gemtuzumab ozogamicin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of CMA-676 in treating patients with acute myeloid leukemia in first relapse.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the efficacy of CMA-676 in terms of the number of patients with acute myeloid leukemia attaining a complete remission. II. Assess the safety of CMA-676 in this patient population.

OUTLINE: This is an open label, single arm, multicenter study. Patients receive CMA-676 IV over 2 hours on day 1. Patients may receive 1 additional dose of therapy 15 to 28 days later. Patients who achieve complete or morphologic remission are followed for an additional 6 months and every 3-6 months thereafter until relapse and/or death.

PROJECTED ACCRUAL: 55 evaluable patients will be accrued. Enrollment will then be extended for up to an additional 55 patients.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically diagnosed CD33 positive acute myeloid leukemia (AML) in first relapse At least 6 months of complete remission No CNS leukemia No AML secondary to exposure to chemotherapy or toxins

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC less than 30,000/mm3 at time of CMA-676 administration Hepatic: Bilirubin no greater than 1.5 mg/dL Renal: Creatinine no greater than 2.0 mg/dL Cardiovascular: No severe cardiac disease Pulmonary: No severe pulmonary disease Other: Not pregnant or nursing Fertile patients must use an effective method of contraception Not known to be HIV positive No prior myelodysplastic syndrome No other active malignancy No uncontrolled infections Able to obtain bone marrow aspirate

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior bone marrow transplantation No prior anti-CD33 antibody therapy Chemotherapy: No prior chemotherapy for AML in first relapse except hydroxyurea At least 24 hours since prior hydroxyurea Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Not specified Other: At least 4 weeks since prior investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 1997-02; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Stanley Berger, MD, Study Chair — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (13):
- United States (13):
  - Arizona Cancer Center, Tucson, Arizona
  - Beckman Research Institute, City of Hope, Duarte, California
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Marlene & Stewart Greenebaum Cancer Center, University of Maryland, Baltimore, Maryland
  - New England Medical Center Hospital, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - New York Presbyterian Hospital - Cornell Campus, New York, New York
  - University of Pennsylvania Cancer Center, Philadelphia, Pennsylvania
  - University of Texas - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Background] Lang K, Menzin J, Earle CC, Mallick R. Outcomes in patients treated with gemtuzumab ozogamicin for relapsed acute myelogenous leukemia. Am J Health Syst Pharm. 2002 May 15;59(10):941-8. doi: 10.1093/ajhp/59.10.941. PMID 12040733
- [Derived] Hibma J, Knight B. Population Pharmacokinetic Modeling of Gemtuzumab Ozogamicin in Adult Patients with Acute Myeloid Leukemia. Clin Pharmacokinet. 2019 Mar;58(3):335-347. doi: 10.1007/s40262-018-0699-5. PMID 30062662